CLINICAL TRIAL: NCT01219296
Title: Retrospective Database Studies From Reproductive Endocrinology Practice Looking at Relationships Between Demographics, Stimulation Protocols and Outcomes, Retrieval and Transfer Outcomes, Number and Quality of Oocytes and Embryos Retrieved and Transferred, Pregnancy Rates and Pregnancy Outcomes.
Brief Title: Retrospective Database Studies
Status: Completed | Type: Observational
Sponsor: Reproductive Medicine Associates of New Jersey (Other)
Responsible Party: Sponsor
Other Study IDs: RMA-00-01
Record Dates: First submitted 2010-10-08; First posted 2010-10-13 (Estimated); Last update posted 2015-11-17 (Estimated); Status verified 2015-11

CONDITIONS: All Patients Undergoing Infertility Treatment
Keywords: infertility; IVF
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

SUMMARY:
Data collection and comparison of relationships between patient demographics, stimulation protocols and outcomes, retrieval and transfer outcomes, number and quality of oocytes and embryos retrieved and transferred, pregnancy rates and pregnancy outcomes.

DETAILED DESCRIPTION:
No patient treatment is associated with the study.

ELIGIBILITY:
Inclusion Criteria:

none

Exclusion Criteria:

none

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients undergoing infertility treatment in our practice.
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2002-06; Primary Completion 2015-10 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Improving Rates while Decreasing Adverse Outcomes | duration of study
  Retrospective database analysis in order to advance the field of reproductive endocrinology, to learn about reproductive aging and diminished ovarian reserve, to correlate oocyte and embryo quality with pregnancy rates and outcomes, and to reduce adverse outcomes such as Ovarian Hyperstimulation Syndrome (OHSS) and multiple pregnancy rates.

CONTACTS AND LOCATIONS:
Overall Officials: Richard T Scott, MD, Principal Investigator — Reproductive Medicine Associates of New Jersey
Locations (1):
- Reproductive Medicine Associates of New Jersey, Basking Ridge, New Jersey, United States